CLINICAL TRIAL: NCT04340661
Title: Effects of a Food Supplement Composed by BIOintestil ® (Bionocol®) on Microbiota and Inflammatory Profile in Irritable Bowel Syndrome Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Targeting Gut Disease S.R.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TGD-01
Record Dates: First submitted 2019-09-03; First posted 2020-04-09 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2020-04

CONDITIONS: Irritable Bowel Syndrome
Keywords: Microbiota; immune system
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bionocol arm (Experimental)
  Interventions: Dietary Supplement: BIOintestil
- Placebo arm (Placebo Comparator)
  Interventions: Dietary Supplement: PLACEBO

INTERVENTIONS:
Dietary Supplement: BIOintestil — Ginger ryzoma powder and Palmrose essential oil (Cymbopogon Martinii)
  Other Names: BIONOCOL
  Arms: Bionocol arm
Dietary Supplement: PLACEBO — Cornstarch
  Arms: Placebo arm

SUMMARY:
The aim of this double blind placebo-controlled study is to evaluate the effect of BIOintestil on fecal microbiota, inflammatory chemokines and symptoms in patients affected by Irritable Bowel Syndrome (IBS).

DETAILED DESCRIPTION:
BIOintestil is a dietary supplement based on Palmrose oil (Cymbopogon martinii) and ginger ryzoma powder. Palmrose oil effects were already established in animal model of colitis and in a pilot study on patients with IBS. In this study, 108 patients will be randomized to receive BIOintestil or placebo in a 1:1 ratio, for four weeks. Fecal and blood samples will be collected at each visit for microbiota and chemokine analysis, patients syntoms will be evaluated by administration of the validated IBS-VAS.

ELIGIBILITY:
Inclusion Criteria:

* willing of sign written informed consent;
* participants affected with Irritable bowel syndrome (IBS) who satisfy Rome III criterias for diagnosis
* body weight between 48 and 104 kg, with a BMI less than 27
* age between 18 and 65 years old

Exclusion Criteria:

* participants that have not taken following medications within 30 days before randomization: steroidal anti-inflammatory drugs, antibiotics or supplemntes or functional foods that may contain probiotics or prebiotics
* women who suspect to be/are pregnant or in lactacy
* participants with Inflammatory bowel disease disgnosis or celiac disease or severe systemic disease
* participants who are intolerant to lactose or with food allergies confirmed
* particpiants with confirmed or suspected hypersensibility to one or more of Bionocol® components
* participants with severe concomitants disease that, by investigator's opinion, interfere with study partecipation
* participants under anticoagulant therapy or with coagulation disease
* participants with renal and hepatic failure
* participants who have taken any investigational drug within 2 month the randomization visit

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2018-12-05 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Changes in fecal Microbiota composition | 4 weeks
  relative abundance of bacteroidetes

SECONDARY OUTCOMES:
Changes in circulating cytokines and chemokines | 4 weeks
  IL-1β, IL-4, IL-6, IL-10,IL-17A,IL-17F, IL-21, IL-22, IL-23, IL-25, IL31, IL-33, IFN-γ, MIP-1b , MCP-1 cytokines and chemokines will be evaluated
Irritable Bowel Syndrome-Visual Analogue Scale (IBS-VAS) score improvement | 4 weeks
  Irritable Bowel Syndrome-Visual Analogue Scale is designed to measure the treatment response of symptoms and well-being in patients suffering from IBS. It is composed by 4 items:
  1) abdominal pain, 2) Abnominal bloating, 3) Satisfaction of the intestinal habits 4) influence on daily life. The patients are asked to record in the VAS-IBS the overall severity of each of the 4 items on a 100-mm-long horizontal line ("very severe discomfort 0" to "no discomfort at all 100").

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Rizzello, MD, Principal Investigator — A.O.U Policlinico S.Orsola-Malpighi
Locations (1):
- A.O.U Policlinico S.Orsola-Malpighi, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No